CLINICAL TRIAL: NCT04880616
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of NBI-827104 in Subjects With Essential Tremor
Brief Title: Safety, Efficacy, and Tolerability of NBI-827104 for the Treatment of Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-827104-ET2016; 2020-006012-24 (EudraCT Number)
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Essential Tremor
Keywords: Movement disorder; Tremor syndrome
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): In treatment period 1 participants will receive increasing doses of NBI-827104 for 28 days. After a 14-day washout period, participants will receive matching placebo for 28 days in treatment period 2.
  Interventions: Drug: NBI-827104; Drug: Placebo
- Sequence 2 (Experimental): In treatment period 1 participants will receive matching placebo for 28 days. After a 14-day washout period, participants will receive increasing doses of NBI-827104 for 28 days in treatment period 2.
  Interventions: Drug: NBI-827104; Drug: Placebo

INTERVENTIONS:
Drug: NBI-827104 — Capsules for oral administration
Drug: Placebo — Capsules matching NBI-827104 for oral administration

SUMMARY:
The main objective of this study is to evaluate the efficacy, safety, and tolerability of NBI-827104 in adults with essential tremor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 to 75 years of age, inclusive at screening.
2. Body mass index (BMI) between 18 and 35 kg/m², inclusive, at screening.
3. Diagnosis of Essential Tremor (inclusive of Essential Tremor plus) as defined by the Movement Disorders Society Consensus Criteria for Tremor.
4. Confirmation of bilateral upper limb action tremor in the absence of overt dystonia, ataxia, or parkinsonism.
5. History of onset of tremor before 65 years of age.
6. Tremor Performance score of ≥ 2 on at least 2 of the 6 upper limb manoeuvres (Item 4) on the TETRAS Performance Subscale and a total TETRAS Performance score ≥15 at screening.
7. All women of childbearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception for at least 90 days after their last dose of study drug.

Exclusion Criteria:

1. Evidence of any acute (at screening or prior to first dose) or chronic disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator.
2. Have direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor.
3. Have known history of other medical or neurological conditions that may cause or explain subject's tremor.
4. Have had prior magnetic resonance guided focused ultrasound or surgical intervention (e.g., deep brain stimulation, ablative thalamotomy or gamma knife thalamotomy).
5. Have a history or evidence of clinically significant cardiac conduction abnormality, uncontrolled bradyarrhythmia, heart failure, or long QT syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Day 28 of Each Treatment Period in Amplitude at Peak Frequency of Postural Tremor | Baseline and Day 28 of each treatment period

SECONDARY OUTCOMES:
Change from Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Performance Score | Baseline up to Day 28 of each treatment period
Change from Baseline in TETRAS Activities of Daily Living (ADL) Score | Baseline up to Day 28 of each treatment period
Clinical Global Impression of Change (CGI-C) | Up to Day 28 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (1):
- Neurocrine Clinical Site, Leiden, CL, Netherlands

IPD SHARING:
Plan to Share IPD: No